CLINICAL TRIAL: NCT04572919
Title: Lateral Advancement Adipo-Fascio-Cutaneous Flap Versus Classic Limberg Flap in The Treatment Of Non-Complicated Pilonidal Sinus: A Prospective Randomized Controlled Trial
Brief Title: Lateral Advancement Flap Versus Classic Limberg Flap in The Treatment Of NonComplicated Pilonidal Sinus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed I Farid, associate professor of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIFarid
Record Dates: First submitted 2020-09-19; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Patients were randomly assigned to undergo lateral advancement flap
  Interventions: Procedure: lateral advancement flap
- group B (Active Comparator): Patients were randomly assigned to undergo classic Limberg flap
  Interventions: Procedure: classic Limberg flap

INTERVENTIONS:
Procedure: lateral advancement flap — Patients were randomly assigned to undergo either lateral advancement flap or classic Limberg flap for treatment of non-complicated pilonidal sinus
  Arms: group A
Procedure: classic Limberg flap — Patients were randomly assigned to undergo either lateral advancement flap or classic Limberg flap for treatment of non-complicated pilonidal sinus
  Arms: group B

SUMMARY:
Background The flaps closure including natal cleft obliteration and eccentric closure are becoming more popular due to their lower rate of recurrence including both the lateral advancement adipo-fascio-cutaneous flap and the classic limberg flap.

Objective This study was aim to compare the results of the surgery for non-complicated pilonidal sinus with the lateral advancement adipo-fascio-cutaneous flap versus the classic Limberg flap.

Patients and methods This study was a prospective randomized controlled, and was conducted on patients with non-complicated pilonidal sinus attending Zagazig University Hospitals, Egypt during the period from February 2017 to August 2019. Patients were randomly assigned to undergo either lateral advancement flap or classic Limberg flap groups. The follow-up period ranged from 12 to 36 months. Patient satisfaction, complications and recurrence rates were analyzed and compared.

DETAILED DESCRIPTION:
Hodges was the first to use the term "pilonidal" (which was derived from the Latin pilus=hair and nidus=nest) in 1988.

The pilonidal disease is usually predisposed by the presence of a deep natal cleft containing a lot of hairs within it, which is also supplies a good environment for maceration, sweating, hairs penetration, and bacterial contamination . A lot of surgical treatment techniques are described for pilonidal sinus disease as simple excision and packing, excision with primary midline closure, marsupialization and eccentric closure by different types of flaps.

Though no surgical technique has been widely accepted, but the flaps closure including natal cleft obliteration and eccentric closure are becoming more popular due to their lower rate of recurrence.

Although the off-midline approach seems optimal for closure, the standard off-midline surgery has not yet been concluded.

According to our best knowledge, no randomized study has yet compared the lateral advancement adipo-fascio-cutaneous flap and the classic Limberg flap. Therefore, the aim of the present study was to compare in a randomized controlled trial the short-term results of the surgical treatment of non-complicated pilonidal sinus with the lateral advancement adipo-fascio-cutaneous flap versus the classic Limberg flap.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-complicated pilonidal sinus
* whose ages ranged from 18 to 60years

Exclusion Criteria:

* elderly patients with comorbid diseases
* scars from a previous pilonidal surgery or recurrent cases
* abscess presentations
* diabetes mellitus, immunodeficiency, or other co-morbidity
* American Society of Anesthesiologists physical status classification grade III-IV
* age < 18years or > 60 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
recurrence | 12 - 36 months
  number of patients recurrence

CONTACTS AND LOCATIONS:
Overall Officials: mohamed farid, MD, Principal Investigator — zagazig university hospital
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
the Study Protocol and the Clinical Study Report are planned to be shared